CLINICAL TRIAL: NCT03532204
Title: Oligometastases of the LIVer Treated With Chemotherapy With ou Without Extracranial Stereotactic Body Radiation Therapy in Patients With Colorectal Cancer
Acronym: OLIVER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0107/1602; NCT03296839 (obsolete NCT alias)
Record Dates: First submitted 2018-01-25; First posted 2018-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Liver Metastases; Colorectal Cancer
Keywords: Oligometastatis; SBRT
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy + SBRT (Experimental): Patients will received 2 courses of chemotherapy before SBRT if no hepatic or extra-hepatic progression identified.
  All liver metastases will be irradiated. 4 doses prescription are allowed (according to the center, and the technique uded and the dosimetric constraints): 3x15 Gy, 4 x 15 Gy, 5 x10 Gy or 5 x 8 Gy.
  The remaining courses of chemotherapy 2 to 3 weeks after completion of SBRT will be administered
  Interventions: Radiation: SBRT; Drug: Chemotherapy
- Chemotherapy (Active Comparator): Patients will receive chemotherapy as initially scheduled
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Radiation: SBRT — Patients will received 2 courses of chemotherapy before SBRT if no hepatic or extra-hepatic progression identified.
  All liver metastases will be irradiated. 4 doses prescription are allowed (according to the center, and the technique uded and the dosimetric constraints): 3x15 Gy, 4 x 15 Gy, 5 x10 Gy or 5 x 8 Gy.
  The remaining courses of chemotherapy 2 to 3 weeks after completion of SBRT will be administered
  Arms: Chemotherapy + SBRT
Drug: Chemotherapy — At investigator's discretion

SUMMARY:
The role of radiotherapy in metastatic cancer has historically been limited to palliation while metastasectomy or radiofrequency has emerged as playing a major role in disease control. Although resection is the standard of care for liver metastasis, 80-90% of patients are not resectable at diagnosis in particular because of the presence of oligometastases. Factors that favour a truly oligometastatic state include a long latent interval between the treatment of the primary tumor and the appearance of metastases.

Oligometastatic cancer is a very heterogeneous disease with respect to several factors including the location of the primary tumor. With the advent of extracranial stereotactic body radiation therapy (SBRT), higher biological equivalent doses can be safely delivered in 3 to 5 fractions, thus potentially ablating all the tissue in the treated area while protecting more efficiently the hosting organ and healthy tissues surrounding the tumors.

In patients with liver oligometastases, in-field local control rates at 2 years range from 70% to 90% with less than 5% severe grade 3 or higher toxicity rates. Retrospective studies indicate that roughly 20% of the patients remain disease-free 2 to 4 years after SBRT.

For patients treated with SBRT some authors found that half of the patients had either no metastatic progression or very little progression in terms of number and site of metastases. The patterns of failure after SBRT for oligometastases in one organ showed that 73% of patients eventually developed new metastases with higher than 80% occurring as new metastases in the same index organ. These findings support the idea of an oligometastatic state in which aggressive local therapy could improve progression-free survival (PFS).

With this phase III study, we sought to evaluate the impact of SBRT on PFS at 2 years in patients with synchronous or metachronous liver-only oligometastases from colorectal cancers patients after a first line chemotherapy for metastatic disease but not having progressed during first line chemotherapy and up to 1 year

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with age ≥18 years and <85 years;
2. Patient with histologically proven colorectal cancer;
3. Patient with a curative surgical treatment (R0) of the primary tumor performed;
4. Oligometastatic disease defined as 1 to 3 liver-only metastases (measurable lesion as per RECIST 1.1);
5. Patient unfit for surgery or with unresectable metastases;
6. Maximal diameter of largest metastasis: 30 mm;
7. Patient naïve of chemotherapy in the metastatic setting or after a first-line of chemotherapy for metastatic disease but not having progressed up to 1 year (i.e. slowly progressing disease);
8. WHO status 0-1;
9. Adequate liver function: bilirubin <3 mg/dL, albumin >2.5 g/dL;
10. Adequate hematological function: absolute neutrophil count (ANC) >1.5 x 10⁹/L; platelets >100 x 10⁹/L, hemoglobin (Hb) >9 g/dL;
11. Normal PT (>70%) and PTT except if the patient uses anticoagulants;
12. Liver enzymes <3 times upper limit of normal;
13. Renal function must be adequate for infusion of iv. contrast agent for CT-scan according to the local policy;
14. Woman of childbearing potential and male patients must agree to use adequate contraception for the duration of study and up to 3 months following completion of therapy;
15. Patient who have received the information sheet, dated and signed the informed consent form;
16. Affiliated to the social security system.

Exclusion Criteria:

1. Healthy liver volume<700 mL
2. Life expectancy <3 months;
3. Patient fit for metastasectomy or hepatectomy;
4. Extrahepatic metastases;
5. Cirrhosis with Child Pugh score B or C;
6. More than one line of chemotherapy in the metastatic setting or rapidly progressing disease;
7. Previous local treatment of liver metastases;
8. Treatment with any other investigational agent against cancer;
9. Malignancies other than mCRC within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, and ductal carcinoma in situ treated surgically with curative intent;
10. Pregnant woman or breast feeding mother;
11. Patient deprived of liberty or placed under the authority of a tutor. Patient with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial. Patient unable to understand the purpose of the study (language, etc.).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-15 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 1 year
  To evaluate the impact of SBRT on Progression-Free Survival (PFS) at 1 year according to RECIST 1.1

SECONDARY OUTCOMES:
Local Control rate | 1 and 3 years
  Defined as the time from the date of randomization to the date of a documented loco-regional event
Overall survival | 3 years
  Defined as the time from the date of randomization to the date of documented death of any cause
Cancer specific survival | 3 years
  Defined as the time from the date of randomization to the date of documented death from cancer or complication from treatment
CTCAE Toxicity Assessment | up to 24 weeks
  Acute/ late toxicity will be assessed according to the flowchart and performed based on CTCAE V4
Quality of life EORTC QLQ C30 | up to 24 weeks
  Will be assessed using self-administered questionnaires EORTC QLQ C30
Quality of life EORTC QLQ CR29 | up to 24 weeks
  Will be assessed using self-administered questionnaire QLQ CR29

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie SERVAGI, MD, Principal Investigator — INSTITUT JEAN GODINOT, REIMS; Gilles CREHANGE, MD, Principal Investigator — CENTRE GEORGES FRANCOIS LECLERC, DIJON